CLINICAL TRIAL: NCT04576260
Title: Effect of a Cognitive Behavioural Therapy Intervention to Improve Sleep on Wellbeing, Dietary Intake and Food Preference: a Feasibility Study.
Brief Title: Effect of CBT Intervention to Improve Sleep on Wellbeing, Dietary Intake and Food Preference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Professor Jason Gill, Professor, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200190177
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Sleep; Diet; Well Being
Keywords: Sleep Extension; Sleep deprivation; Dietary intake; Well being; Cognitive Behavioural Therapy; Cognitive Behavioural Therapy for Insomnia; CBTi; Sleep Quality
MeSH Terms: conditions — Sleep Deprivation; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial with two groups CBT intervention group and control group.
Who Masked: Outcomes Assessor
Masking Description: Members of the research team that perform measurements are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I Group (Experimental): Participants in the CBT-I group will undertake weekly sessions for a duration of 8 weeks with a trained psychologist through Zoom or Skype Calls.
  Interventions: Behavioral: Cognitive Behavioural Therapy for Insomnia
- Control group (No Intervention): The control group will be asked to maintain the usual lifestyle for the duration of the study

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Insomnia — Weekly CBTI training
  Arms: CBT-I Group

SUMMARY:
The study aims to investigate the effects of Cognitive Behavioural therapy intervention on sleep and it's effects on well-being, dietary intake and food preferences during COVID-19. The study will investigate whether delivery of a CBT intervention will lead to an improvement in sleep quality and sleep duration and will consequently improve metabolic health. The participants will be randomized into two groups with one half in the intervention arm and the other in the control arm of the study.

DETAILED DESCRIPTION:
Reduced sleep duration and sleep quality have become increasingly important areas in the study and epidemiology of sleep and are linked with numerous health risks. The Centers for Disease Control and Prevention have found that in the last few years there has been a significant reduction in sleep duration in adults, with an average duration of <7 hours, with some suggestion that this can contribute to increased risk of obesity and type 2 diabetes.

Studies on sleep restriction have observed that even a single night of sleep deprivation leads to a reduction in insulin sensitivity and increases the prevalence of diabetes. Similarly shortened and/or poor-quality sleep has been found to cause dysregulation in ghrelin and leptin levels, which can increase energy intake and motivation to seek out foods with higher fat and sugar content. Although a wide range of research focuses on the effects of short sleep and its impact on health, few studies have focused on whether improving sleep can improve cardiometabolic outcomes.

Research has estimated that almost 30% of individuals suffer from insomnia or insomnia like symptoms. The most common method to combat this has been over-the-counter medication and hypnotics; however, there is very little evidence available on the efficacy of such treatments. Over the years, Cognitive Behavioural Therapy has been found to produce long term and significant results in individuals with insomnia. It has shown to significantly improve the various parameters of sleep such as sleep latency, wake after sleep onset, sleep efficiency and sleep quality. Studies on patients with primary insomnia have shown that those undergoing CBT treatment improve their sleep by an average of 6 hours and improve their sleep efficiency. Furthermore, those undergoing CBT have shown long term improvements with healthy circadian rhythms, regulated hormonal secretory patterns and blood glucose levels.

A research study on short sleep duration with an intervention consisting of behavioural consultations focusing on extending sleep found that extending sleep, through this intervention, reduced the intake of free sugars, fat, and carbohydrates. Since CBT requires minimal intervention, it could be considered as the ideal mode of therapy to improve sleep.

In the current scenario, with the significant effects of COVID-19 observed on morbidity, daily lifestyle behaviours, and mental health, an effective psychological intervention may help to improve both mental and physiological health. This study aims to investigate the effects of an intervention which improves sleep on metabolic health outcomes. Through this study, the investigators aim to test the feasibility of a CBT intervention in improving sleep in our target population consisting of overweight/obese adults reporting poor sleep and to further understand participants' experiences with the CBT to improve health and sleep outcomes during a pandemic.

The study is a randomized control trial where all participants will undergo the screening and baseline measurements. On completion of these procedures, the participants in the intervention group will undergo an 8-week session plan for 1 hour every week conducted online by a certified CBT-i trained psychologist. On completion of the study, all participants will be asked to undertake post-intervention measures.

ELIGIBILITY:
Inclusion Criteria:

* BMI above 25kg/m2.
* Self-reported sleep of <7hrs (confirmed through actigraphy).
* A global score of >5 on the Pittsburgh Sleep Quality Index (PSQI)
* Participants on any kind of self-prescribed or over the counter medication for sleep, will be included in the study after a two-week interval for elimination drug from the system.

Exclusion Criteria:

* Presence of sleep-related disorders measured through the Sleep Disorder Symptoms Checklist (SDSCL-25)
* Any serious medical conditions which might influence sleep i.e. cardiovascular diseases, diabetes, cancer, respiratory disease, other than mild asthma.
* History of bariatric surgery.
* Taking any kind of prescribed hypnotics or sleep medication
* Taking any kind of medication which might affect appetite
* Participating in any kind of dietary and/or weight loss programs
* Taking Antidepressants
* Substance or alcohol abuse
* Shift work
* Currently having to wake up at night to care for another person
* Suffering from and/or receiving treatment for a mental health conditions or sleep apnea.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Sleep Duration | 0-12 weeks
  Change in accelerometer measured total sleep time

SECONDARY OUTCOMES:
Sleep Efficiency | 0-12 weeks
  Changes in Accelerometer measured sleep efficiency
Sleep Latency | 0-12 weeks
  Changes in Accelerometer measured sleep latency
Total Sleep Time | 0-12 weeks
  Changes in Accelerometer measured Total sleep Time
Total Time in Bed | 0-12 weeks
  Changes in Accelerometer measured Total time in bed
Wake After Sleep Onset | 0-12 weeks
  Changes in Accelerometer measured Wake after sleep onset
Subjective Sleep Quality | 0-12 weeks
  Changes in subjective sleep quality measured by The Pittsburgh Sleep Quality Index
Sleep Disturbances | 0-12 weeks
  Changes in sleep disturbances measured by The Pittsburgh Sleep Quality Index
Use of Sleeping Medication | 0-12 weeks
  Changes in use of sleeping medication measured by The Pittsburgh Sleep Quality Index
Daytime Dysfunction | 0-12 weeks
  Changes in daytime dysfunction measured by The Pittsburgh Sleep Quality Index
Habitual Sleep Efficiency | 0-12 weeks
  Changes in habitual sleep efficiency measured by The Pittsburgh Sleep Quality Index
Sleep Duration (self-reported) | 0-12 weeks
  Changes in sleep duration measured by The Pittsburgh Sleep Quality Index
Excessive Daytime Sleepiness | 0-12 weeks
  Changes in excessive daytime sleepiness measured by the Epworth Sleepiness Scale
  Scale range:
  Would never nod off 0 Slight chance of nodding off 1 Moderate chance of nodding off 2 High chance of nodding off 3
  Scoring Interpretation:
  Minumum score is 0 and maximum score is 24. 0-5 - Lower Normal Daytime Sleepiness 6-10 - Higher Normal Daytime Sleepiness 11-12 - Mild Excessive Daytime Sleepiness 13-15 - Moderate Excessive Daytime Sleepiness 16-24 - Severe Excessive Daytime Sleepiness
Mental Well-being | 0-12 weeks
  Changes in cognitive, affective and social dimensions of mental health measured by the Warwick-Edinburgh Mental Well-being Scale
  Scale range:
  None of the time 1 Rarely 2 Some of the time 3 Often 4 All of the time 5
  Scoring Interpretation:
  The minimum score is 14 and maximum score is 70. The higher the scores indicate a greater positive mental wellbeing.
Depression | 0-12 weeks
  Changes in depressive symptoms measured by the Patient Health Questionnaire-9
  Scale range:
  Not at all 0 Several days 1 More than half the days 2 Nearly every day 3
  Scoring Interpretation:
  The minimum score is 0 and maximum score is 20. 0-5 - mild 6-10 - moderate 11-15 - moderately severe 16-20 - severe depression
Anxiety | 0-12 weeks
  Changes in anxiety measured by the Generalized Anxiety Disorder-7
  Scale range:
  Not at all 0 Several days 1 More than half the days 2 Nearly every day 3
  Scoring Interpretation:
  The minimum score is 0 and maximum score is 21. 0-5 mild 6-10 moderate 11-15 moderately severe anxiety 15-21 severe anxiety.
Food preference | 0-12 weeks
  Changes in explicit liking and explicit wanting measured by the Leeds Food Preference Questionnaire
  Scale range:
  The computerized asessment includes a 100mm visual analogue scale and at the end of the response item participants will be asked: "How much do you want some of this food now?
  Scoring:
  The minimum score for VAS scale is 0 and maximum is 100. Scores are recorded and converted in to mean scores for high fat, low fat, sweet or savoury food types and different fat-taste combinations.
Food reward | 0-12 weeks
  Changes in implicit wanting and food choice measured by the Leeds Food Preference Questionnaire
  Scale range:
  The computerized asessment where participants are presented with two images and they choose which they like.
  Scoring:
  Reaction time for each answer is recorded and converted in to mean scores for high fat, low fat, sweet or savoury food types and different fat-taste combinations.
Food cravings | 0-12 weeks
  Changes in craving control, craving for sweet, craving for savoury and positive mood measured by the Control of Eating Questionnaire
  Scale range:
  The asessment includes a 20 items with a 10 point scale ranging from "not at all" to "extremely" and 1 item with free text answer.
  Scoring:
  The minimum score for VAS scale is 0 and maximum is 100. The sum of items were calculated and divide by number of items in the subscale. Higher the score indicates higher cravings. Positive mood subscales and Craving Control subscales the scores were reversed, so great score indicated greater level of positve mood and craving control.
Dietary Intake | 0-12 weeks
  Changes in 24 hour food recall measured by the Myfood24 food diary

OTHER OUTCOMES:
Anthropometric Measures | 0-12 weeks
  Changes in self reported weight
Anthropometric measures | 0-12 weeks
  Changes in self reported BMI
Participant Interviews | 0-12 weeks
  Participant feedback and information provided through interviews

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gill, PhD, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom